CLINICAL TRIAL: NCT03747549
Title: Acupuncture for Insertional Achilles Tendinopathy in the Primary Care Setting: a Randomized Comparative Effectiveness Trial
Brief Title: Acupuncture for Insertional Achilles Tendinopathy Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FWH20180170H
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insertional Achilles Tendinopathy
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture and Home Exercise (Experimental): Acupuncture and home exercise.
  Interventions: Other: Acupuncture and Home Exercise
- Home Exercise Alone (Active Comparator): The prescribed home exercise program alone.
  Interventions: Other: Home Exercise Alone

INTERVENTIONS:
Other: Acupuncture and Home Exercise — Acupuncture (needles will be placed at BL 60, BL 61, KI 3, KI 4 with needles directed into the Achilles tendon. Needles inserted until a firm catch of the needle entering the tendon was appreciated. Energy (a small electrical current) is placed from KI 3(-) KI 4(+) and BL 61 (-) BL 60(+) at 30 Hz for 15min) plus the prescribed home exercise program
  Arms: Acupuncture and Home Exercise
Other: Home Exercise Alone — The prescribed home exercise program alone.
  Arms: Home Exercise Alone

SUMMARY:
The purpose of this study is to compare acupuncture plus a prescribed home exercise program versus a prescribed home exercise program alone to determine which has better outcomes at improving pain relief and physical function in adult patients with insertional Achilles tendinopathy.

The investigators want to compare a combination of two standard of care treatments (acupuncture plus a prescribed home exercise program) versus a single standard of care treatment (a prescribed home exercise program) to determine which has better outcomes with improving pain relief and physical function in patients with insertional Achilles tendinopathy. The investigators hypothesize that there will be a significant improvement in pain and functional outcomes, both acutely and over time, in the acupuncture plus a prescribed home exercise program group versus the group performing a prescribed home exercise program alone. The investigators will measure Achilles pain relief and physical function immediately prior to treatment (baseline), immediately after the initial treatment at day 1, 2 weeks, 4 weeks, 6 weeks, and 12 weeks using the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A). After 3 months, patients with continuing pain in the non-acupuncture arm will be given the option to crossover to the acupuncture arm of the study for an additional 12 weeks of treatment with the subject's concurrence.

DETAILED DESCRIPTION:
Screening Visit (research-related):

* Obtain and document signed Informed Consent document and HIPAA Authorization.
* Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria including previous encounter, vital signs review, co-morbidities, demographics, and problems list.
* Record: Date of birth, age, gender, race, ethnicity, DoD ID number, name of standard of care medications (over-the-counter and prescription), current email address (to be used for scheduling), height (in inches), weight (in pounds),history of prior injury to the injured leg, and note any prior acupuncture received for Achilles tendinopathy.
* If the subject is an active duty member, the investigators will ask: Have you or are you currently on a fitness restriction for Achilles tendinopathy.

If so, what are/were the dates of the restriction?

• There are several standard of care treatments for Achilles tendinopathy which include physical therapy as well as a prescribed home exercise program. The investigators will standardize what patients in this study are receiving by having all subjects follow a standard home exercise program defined as the Insertional Achilles Tendinopathy Eccentric Training Protocol and have them discontinue any formal physical therapy or other therapies when entering this study. Regular physical activity such as exercise is allowed.

Randomization: Subjects will be randomized into 1 of 2 research treatment groups using block randomization with repeated measures:

* Group 1: Acupuncture (needles will be placed at BL 60, BL 61, KI 3, KI 4 with needles directed into the Achilles tendon. Needles inserted until a firm catch of the needle entering the tendon was appreciated. Energy (a small electrical current) is placed from KI 3(-) KI 4(+) and BL 61 (-) BL 60(+) at 30 Hz for 15min) plus the prescribed home exercise program
* Group 2: The prescribed home exercise program alone.

Visit 1-Day 1 (may be same day as screening visit) (research-related)::

* Subjects will be given a study diary to document the number of times they performed the Insertional Achilles Tendinopathy Eccentric Training Protocol.
* Subjects will be advised to complete exercises twice a day for three sets of 15 repetitions for 12 weeks.4
* Administer the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A)
* Document Morphine Equivalent Units (MEU) and over-the-counter and prescription medications used in the last 2 weeks.
* Self-reported pain severity pre-intervention (0 for no pain to 10 being the worst pain)
* Research treatment intervention according to their randomization group:

Group 1:

Subjects will be asked what their expectations are regarding acupuncture's effectiveness for Achilles tendinopathy.

The prescribed home exercise program will be reviewed. Acupuncture will be performed. Research coordinator will record the name of the investigator performing the acupuncture

Group 2:

The prescribed home exercise program will be reviewed. Self-reported pain severity post-intervention (0 for no pain to 10 being the worst pain)

Visit 2-Week 2 (research-related)::

* Subjects' study diaries will be reviewed and the number of times the Insertional Achilles Tendinopathy Eccentric Training Protocol was performed will be documented.
* Subjects will be reminded to complete the exercises twice a day for three sets of 15 repetitions for 12 weeks.
* Administer the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A)
* Document Morphine Equivalent Units (MEU) and over-the-counter and prescription medications used since the last visit.
* Self-reported pain severity pre-intervention (0 for no pain to 10 being the worst pain)
* Research treatment intervention according to their randomization group:

Group 1:

The prescribed home exercise program will be reviewed. Acupuncture will be performed. Research coordinator will record the name of the investigator performing the acupuncture

Group 2:

The prescribed home exercise program will be reviewed. Self-reported pain severity post-intervention (0 for no pain to 10 being the worst pain)

Visit 3-Week 4 (research-related):

* Subjects' study diaries will be reviewed and the number of times the Insertional Achilles Tendinopathy Eccentric Training Protocol was performed will be documented.
* Subjects will be reminded to complete the exercises twice a day for three sets of 15 repetitions for 12 weeks.
* Administer the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A)
* Document Morphine Equivalent Units (MEU) and over-the-counter and prescription medications used since the last visit.
* Self-reported pain severity pre-intervention (0 for no pain to 10 being the worst pain)
* Research treatment intervention according to their randomization group:

Group 1:

The prescribed home exercise program will be reviewed. Acupuncture will be performed. Research coordinator will record the name of the investigator performing the acupuncture

Group 2:

The prescribed home exercise program will be reviewed. Self-reported pain severity post-intervention (0 for no pain to 10 being the worst pain)

Visit 4-Week 6 (research-related)::

Subjects' study diary will be reviewed and the number of times the Insertional Achilles Tendinopathy Eccentric Training Protocol was performed will be documented.

* Subjects will be reminded to complete the exercises twice a day for three sets of 15 repetitions for 12 weeks.4
* Administer the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A)
* Document Morphine Equivalent Units (MEU) and over-the-counter and prescription medications used since the last visit.
* Self-reported pain severity pre-intervention (0 for no pain to 10 being the worst pain)
* Research treatment intervention according to their randomization group:

Group 1:

The prescribed home exercise program will be reviewed. Acupuncture will be performed. Research coordinator will record the name of the investigator performing the acupuncture

Group 2:

The prescribed home exercise program will be reviewed. Self-reported pain severity post-intervention (0 for no pain to 10 being the worst pain)

Visit 5-Week 12 (research-related)::

* Collect subjects' study diaries.
* Administer the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A)
* Document Morphine Equivalent Units (MEU) and over-the-counter and prescription medications used since the last visit.
* Self-reported pain severity (0 for no pain to 10 being the worst pain)
* Ask if subjects' expectations were met or changed regarding acupuncture's effectiveness for Achilles Tendinopathy. (Group 1 ONLY)

CROSSOVER: At Visit 5 (final visit), patients in the non-acupuncture group with continuing pain will be given the option to crossover into the acupuncture arm of the study where they will complete visit 1 through 5. Visit 1 will be on the same day with corresponding measures as described above for a total study enrollment time of 24 weeks.

ELIGIBILITY:
** THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY **

Inclusion Criteria:

* Male and female DoD beneficiaries, age 18 years or older
* diagnosed with Achilles tendinopathy OR patients meeting criteria of pain 2cm or less from the insertion to the Achilles tendon on the calcaneus.
* Patients must have had pain for greater than 8 weeks and a VISA-A score less than 60.

Exclusion Criteria:

* Pregnant
* Active cellulitis over the area of needle insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Change in pain over time as measured by the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A) | the first visit, 2 weeks, 4 weeks, 6 weeks, and 12 weeks
  Change in pain over time as measured by the Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A). The VISA-A is measured as a score out of 100, where a lower score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hawks, MD, Principal Investigator — Mike O'Callaghan Military Medical Center
Locations (2):
- United States (2):
  - 96th Medical Group, Eglin Air Force Base, Florida
  - Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li HY, Hua YH. Achilles Tendinopathy: Current Concepts about the Basic Science and Clinical Treatments. Biomed Res Int. 2016;2016:6492597. doi: 10.1155/2016/6492597. Epub 2016 Nov 3. PMID 27885357
- [Background] Robinson JM, Cook JL, Purdam C, Visentini PJ, Ross J, Maffulli N, Taunton JE, Khan KM; Victorian Institute Of Sport Tendon Study Group. The VISA-A questionnaire: a valid and reliable index of the clinical severity of Achilles tendinopathy. Br J Sports Med. 2001 Oct;35(5):335-41. doi: 10.1136/bjsm.35.5.335. PMID 11579069
- [Background] Iversen JV, Bartels EM, Langberg H. The victorian institute of sports assessment - achilles questionnaire (visa-a) - a reliable tool for measuring achilles tendinopathy. Int J Sports Phys Ther. 2012 Feb;7(1):76-84. PMID 22319681
- [Background] Childress MA, Beutler A. Management of chronic tendon injuries. Am Fam Physician. 2013 Apr 1;87(7):486-90. PMID 23547590
- [Background] Rowe V, Hemmings S, Barton C, Malliaras P, Maffulli N, Morrissey D. Conservative management of midportion Achilles tendinopathy: a mixed methods study, integrating systematic review and clinical reasoning. Sports Med. 2012 Nov 1;42(11):941-67. doi: 10.1007/BF03262305. PMID 23006143
- [Background] Arnold MJ, Moody AL. Common Running Injuries: Evaluation and Management. Am Fam Physician. 2018 Apr 15;97(8):510-516. PMID 29671490
- [Background] Hawks MK. Successful Treatment of Achilles Tendinopathy with Electroacupuncture: Two Cases. Med Acupunct. 2017 Jun 1;29(3):163-165. doi: 10.1089/acu.2017.1232. PMID 28736593
- [Background] Breivik EK, Bjornsson GA, Skovlund E. A comparison of pain rating scales by sampling from clinical trial data. Clin J Pain. 2000 Mar;16(1):22-8. doi: 10.1097/00002508-200003000-00005. PMID 10741815
- [Background] Ludington E, Dexter F. Statistical analysis of total labor pain using the visual analog scale and application to studies of analgesic effectiveness during childbirth. Anesth Analg. 1998 Sep;87(3):723-7. doi: 10.1097/00000539-199809000-00045. No abstract available. PMID 9728862